CLINICAL TRIAL: NCT02268747
Title: Efficacy and Safety of Single Agent Pan-HER Inhibitor Dacomitinib in the Treatment of Locally Advanced Unresectable or Metastatic Squamous Cell Cancer of the Skin or With Clinical Contraindication to Surgery
Brief Title: Efficacy and Safety of Dacomitinib in the Treatment of Skin Squamous Cell Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DACOMINT14; 92/14 (Other: INT)
Record Dates: First submitted 2014-08-09; First posted 2014-10-20 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Skin Squamous Cell Cancer
Keywords: skin squamous cell cancer panHER inhibitor Dacomitinib
MeSH Terms: interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dacomitinib (Experimental): Patients will assume Dacomitinib 30 mg daily for the first 2 weeks. If the highest skin toxicity will be of grade <2, then the patients will start dacomitinib at 45 mg once daily and they will be clinically assessed every cycle (i.e. every 28 days).
  If the highest skin toxicity will be grade >2, then the patient will interrupt the treatment following the criteria for dose reduction.
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — The patients will assume Dacomitinib 30 mg daily for the first 2 weeks. If the highest skin toxicity will be of grade <2, then the patients will start dacomitinib at 45 mg once daily and they will be clinically assessed every cycle (i.e. every 28 days).
  If the highest skin toxicity will be grade >2, then the patient will interrupt the treatment following the criteria for dose reduction.
  Other Names: PF-00299804

SUMMARY:
This is an open label, monocentric, uncontrolled phase II trial with Dacomitinib, a pan-HER inhibitor, in unresectable or metastatic skin SCC.

HER2 expression is common in skin SCC, being reported with high rates, even if in small studies.

Coexpression of EGFR, HER2 and HER3 is present in skin SCCs but not in normal skin and it could be associated with the malignant phenotype. In this frame Dacomitinib could play a role in the increase of the response rate.

DETAILED DESCRIPTION:
The patients will assume Dacomitinib 30 mg daily for the first 2 weeks. If the highest skin toxicity will be of grade <2, then the patients will start dacomitinib at 45 mg once daily and they will be clinically assessed every cycle (i.e. every 28 days).

If the highest skin toxicity will be grade >2, then the patient will interrupt the treatment following the criteria for dose reduction.

Tumor evaluation will be performed at baseline and every other cycle. Response will be assessed according to RECIST 1.1. The patient will continue to assume the study drug until disease progression, unacceptable toxicity or any medical condition that will suggest to stop the treatment for patient's safety

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to treatment
* Histological diagnosis of squamous cell carcinoma of the skin not amenable to surgical treatment with curative purposes or with clinical contraindication to surgery (examples of medical contraindications to surgery include but are not limited to: skin SCC that has recurred in the same location after two or more surgical procedures and curative resection is deemed unlikely; anticipated substantial morbidity and/or deformity from surgery (e.g., removal of all or part of a facial structure, such as nose, ear, eyelid, eye; or requirement for limb amputation); anticipated difficulty in obtaining a curative resection due to the location of the tumour, the size of disease; anticipated difficulty in reconstructing the area that will be surgically removed; significant comorbidities that preclude the feasibility of a radical surgery
* Presence of measurable disease according to RECIST 1.1
* ECOG performance status 0-2
* Age≥ 18 years
* For men and women in the fertile period: the use of birth control systems during treatment

Exclusion Criteria:

* Previous treatment with tyrosine kinase inhibitors or monoclonal antibodies directed against EGFR
* Any toxicity CTC grade> 2 from previous treatments not yet resolved
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Response rate to Dacomitinib | 24 months
  Response rate (partial response, PR + complete response, CR) to Dacomitinib

SECONDARY OUTCOMES:
Compliance to the treatment and safety | 24 months
  Compliance to the treatment and safety
Disease control | 24 months
  Disease control (stable disease (SD) + PR + CR)
PFS and OS | 24 months
  Progression-Free Survival (PFS) and Overall Survival (OS)
Percentage of patients initially not considered for surgery due to difficulty to obtain a curative treatment that undergo surgery after dacomitinib | 24 months
  Percentage of patients initially not considered for surgery due to difficulty to obtain a curative treatment that undergo surgery after dacomitinib

OTHER OUTCOMES:
Analysis of mutational/gene expression | 24 months
  Translational research regarding the analysis of pERK, Ki67, pSTAT3 p27, pEGFR and other mutational/gene expression analysis to be determined within the study period. Correlation of immunohistochemistry analysis of these markers and response to treatment or to onset of acquired resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bossi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Milan, Italy, Italy